CLINICAL TRIAL: NCT04422860
Title: Remineralization Efficacy of Gum Arabic Varnish Versus Fluoride Varnish and CPP-ACP With Fluoride Based Varnish on Initial Carious Lesions. a Randomized Controlled Clinical Trial.
Brief Title: Remineralization Efficacy of Gum Arabic Varnish.
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hesham samaha, Master's Degree Student- Faculty of Dentistry, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEBD-2
Record Dates: First submitted 2020-06-04; First posted 2020-06-09 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-07

CONDITIONS: Caries,Dental; Remineralization; White Spot Lesion
Keywords: Initial carious lesion; Gum Arabic; Remineralization power; fluoride varnish; Mi varnish; Acacia senegal
MeSH Terms: conditions — Dental Caries | interventions — Gum Arabic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Gum Arabic varnish (Experimental): Gum arabic (Acacia senegal) is an exudate obtained from Acacia senegal stems and roots, and other similar African Acacia species. It consists mainly of high molecular weight polysaccharides high concentrations of calcium, magnesium, and potassium salts which can potentially increase tooth remineralization.
  Interventions: Drug: Gum Arabic varnish
- Sodium Fluoride varnish (Active Comparator): The gold standard remineralizing agent recommended by the guidelines.
  Interventions: Drug: Proflourid Varnish,VOCO
- 10% w/v CPP-ACP, 5% sodium fluoride varnish (Active Comparator): CPP-ACP is the most studied non fluoride remineralizing agent.
  Interventions: Drug: MI Varnish,GC Japan Inc.

INTERVENTIONS:
Drug: Gum Arabic varnish — Powdered exudate from various Acacia species, especially A. senegal (Leguminosae).
  Other Names: Acacia senegal
  Arms: Gum Arabic varnish
Drug: Proflourid Varnish,VOCO — 5% NaF varnish
  Arms: Sodium Fluoride varnish
Drug: MI Varnish,GC Japan Inc. — CPP-ACP with fluoride based varnish
  Arms: 10% w/v CPP-ACP, 5% sodium fluoride varnish

SUMMARY:
The aim of this study is to evaluate the remineralizing capacity of Gum Arabic varnish and its implementation into clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients with initial carious lesions.
* Proper Oral hygiene.

Exclusion Criteria:

* Patients with a compromised medical history.
* Patients with active severe periodontal disease.
* Patients with hypoplastic or hypomineralized teeth.

Ages: 17 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
Remineralization through determination of lesion progression or regression | Change from baseline at 3,6, 9 months
  Determination of lesion level by DIAGNOdent which provides a laser fluorescence feedback to give a numerical readout reflects the amount of demineraliztion.

SECONDARY OUTCOMES:
Caries lesion activity assessment | Change from baseline at 3,6, 9 months
  Visual (change in Surface Appearance) - tactile ( change in Tactile Feeling of the surface by an explorer)

CONTACTS AND LOCATIONS:
Overall Officials: Rawda H. A.ElAziz, Post Phd, Study Director — Lecturer at faculty of Dentistry- Cairo University; Rasha R Hassan, Study Chair — Assistant Professor at faculty of Dentistry- Cairo University; Ahmed H. Samaha, BSc, Principal Investigator — Master's Degree student at faculty of Dentistry- Cairo University
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

REFERENCES:
- [Background] Philip N. State of the Art Enamel Remineralization Systems: The Next Frontier in Caries Management. Caries Res. 2019;53(3):284-295. doi: 10.1159/000493031. Epub 2018 Oct 8. PMID 30296788
- [Background] Onishi T, Umemura S, Yanagawa M, Matsumura M, Sasaki Y, Ogasawara T, Ooshima T. Remineralization effects of gum arabic on caries-like enamel lesions. Arch Oral Biol. 2008 Mar;53(3):257-60. doi: 10.1016/j.archoralbio.2007.10.004. Epub 2007 Nov 26. PMID 18036508